CLINICAL TRIAL: NCT06863844
Title: Study for the Evaluation of Molecular Markers Extracted From PRedittivI DNA of Clinical Outcomes and Response to Systemic Therapy in Patients With UROthelial Tumor.
Brief Title: The Evaluation of Molecular Markers From PRedittivI DNA of Clinical Outcomes in Patients With UROthelial Tumor
Acronym: PROCURO
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: PROCURO; RC-2022-2773372 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2025-01-10; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-11

CONDITIONS: Urothelial Neoplasm
Keywords: biomarker

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The genetic characterization of urothelial tumor disease has brought to light important information about the biology of the disease. The evaluation of molecular DNA markers on tumor tissue could be an approach able to provide important information on the possible aggressiveness of the disease and the sensitivity/resistance profile to drugs commonly adopted in the advanced stage. The main objective of this study is to identify specific molecular profiles from DNA capable of predicting the clinical course of the disease and the possible sensitivity/resistance of the disease to systemic treatments

DETAILED DESCRIPTION:
retrospective and prospective evaluation concerning the identification of molecular profiles on DNA obtained from tumor tissue previously obtained from patients with urothelial cancer and analyzed with massive sequencing method (Next Generation Sequencing).

Analysis of data obtained from anamnestic data, clinical data, blood chemistry tests, histopathological examinations and instrumental imaging.

ELIGIBILITY:
Inclusion Criteria For the retrospective part:

- Patients diagnosed with locally advanced operated or metastatic urothelial cancer in follow-up or treatment

Exclusion Criteria For the retrospective part:

- Deceased patients who have not already performed the NGS analysis from clinical practice.

For the prospective part:

Patients

* aged > 18 years
* suffering from locally advanced or metastatic urothelial neoplasia
* with the availability of tumor tissue obtained during surgery on a primary tumor or metastasis or during a diagnostic biopsy.

Patients included in the study will also have to consciously express their willingness to participate in the study after signing the written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with urothelial cancer
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
evaluation of the prognostic and predictive role of response to systemic therapy of specific molecular markers extracted from tumor DNA. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  The study involves the analysis by massive sequencing (Next Generation Sequencing) of molecular profiles of tumor DNA extracted from tumor tissue obtained during surgery (on primary and/or metastases) or diagnostic biopsy performed as part of the normal clinical care pathway. These data will be integrated with information relating to anamnestic data and clinical, laboratory and instrumental parameters of patients with urothelial neoplasia

SECONDARY OUTCOMES:
molecular profiles predictive of response/resistance to chemotherapy, immune-checkpoint inhibitors, target therapy | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Search for molecular profiles predictive of response/resistance to chemotherapy, immune-checkpoint inhibitors, target therapy

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Massari, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero Universitaria Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No